CLINICAL TRIAL: NCT03476018
Title: Z-100 Pharmacological Trial: A Randomised Placebo-controlled Trial of Z-100 Plus Radiation Therapy in Subjects With Locally Advanced Cervical Cancer
Brief Title: Trial to Optimally Show the Pharmacological Action of Z-100
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Z100-02
Record Dates: First submitted 2018-03-04; First posted 2018-03-23 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — specific substance maruyama

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos
- 0.2 microgram Z-100 (Experimental)
  Interventions: Drug: Z-100
- 2 microgram Z-100 (Experimental)
  Interventions: Drug: Z-100
- 20 microgram Z-100 (Experimental)
  Interventions: Drug: Z-100

INTERVENTIONS:
Drug: Z-100 — Twice a week until 29 days after completion of chemoradiotherapy, then once every 14 days
  Arms: 0.2 microgram Z-100; 2 microgram Z-100; 20 microgram Z-100
Drug: Placebos — Twice a week until 29 days after completion of chemoradiotherapy, then once every 14 days
  Arms: Placebo

SUMMARY:
The objective of this clinical trial is to evaluate the change of the immunological parameter levels in FIGO stage IIIB cervical cancer subjects by administration of Z-100

ELIGIBILITY:
Inclusion Criteria:

1. FIGO stage (2008): IIIB, cervical cancer
2. Pathologically confirmed squamous cell carcinoma of the cervix
3. Subjects with treatment-naive cervical cancer
4. Subjects without enlargement (≥15 mm in the short axis) in the lower abdominal para-aortic lymph node
5. Subjects ≥21, ≤79 years of age at informed consent
6. Subjects for whom it is considered possible to carry out intracavitary radiation in radiotherapy
7. Subjects for whom it is considered possible to carry out concurrent cisplatin treatment with radiotherapy
8. Eastern Cooperative Oncology Group Performance Status: 0-2
9. Subjects with the following organ functions; (1) WBC ≥3,000/mm3 (2) Platelet count ≥100,000/mm3 (3) Hemoglobin ≥9.5 g/dL (correction by medication, e.g. blood transfusion, iron compounds, is allowed) (4) Total bilirubin ≤ three (3) times the upper limit of reference value at the clinical testing laboratory (5) AST, ALT ≤ three (3) times the upper limit of reference value at the clinical testing laboratory (6) Creatinine clearance: ≥50 mL/min
10. Subjects who are willing to give informed consent

Exclusion Criteria:

1. Subjects who have a double cancer or are being treated for that
2. Subjects who have suffered from cancers other than cervical cancer within 5 years prior to obtaining consent
3. Subjects with cancer of the cervical stump which is judged by the investigator
4. Subjects who have a history of being diagnosed of autoimmune disease
5. Subjects who have a history of radiotherapy in the pelvis
6. Subjects who have a history of hypersensitivity to cisplatin or other medical agents which contain platinum
7. Subjects complicated with a serious drug allergy
8. Subjects with a serious complication (poorly controlled hypertension, haemorrhagic tendency, connective tissue disease being treated with steroid)
9. Pregnant women, nursing mothers or subjects who desire pregnancy during the trial period
10. Subjects who have ongoing infection of human immunodeficiency virus (HIV), active hepatitis B virus (HBV), hepatitis C virus (HCV)
11. Subjects with symptomatic tuberculosis at the date of obtaining consent
12. Subjects who have received any other investigational medicinal products or medical devices within 28 days prior to obtaining consent
13. Other subjects considered inappropriate to participate in the trial by the investigator

Ages: 21 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change in the number of immunological cells | 2 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Disease-specific survival | 2 years
Recurrence-free survival | 3 years
Rate of adverse events/adverse drug reactions | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Zeria Investrigative Sites, Hanoi
  - Zeria Investigative sites, Ho Chi Minh City